CLINICAL TRIAL: NCT06881017
Title: Establishment of Precision Targeted Therapy Strategies for Advanced Gastric Cancer Based on Novel Molecular Subtyping: an Umbrella Phase II Exploratory Clinical Study
Brief Title: Establishment of Precision Targeted Therapy Strategies for Advanced Gastric Cancer Based on Novel Molecular Subtyping
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: China Medical University, China (Other)
Responsible Party: Principal Investigator, Xiujuan Qu, Director, China Medical University, China
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-GC-II-023
Record Dates: First submitted 2025-03-09; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Gastric Cancer; HER2 + Gastric Cancer; CLDN18.2-positive Adenocarcinoma of the Gastroesophageal Junction; PD-L1 Positive
Keywords: gastric cancer; HER2; CLDN18.2; PD-L1
MeSH Terms: conditions — Stomach Neoplasms | interventions — Trastuzumab; apatinib; S 1 (combination); Capecitabine; Oxaliplatin; zolbetuximab; SHR-1701

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (7):
- Cohort 1 (Experimental): HER2(+)&CLDN18.2(+)&PD-L1(+)
  Interventions: Drug: Trastuzumab; Drug: Adebrelimab; Drug: S-1; Drug: zolbetuximab; Drug: SHR-A1904
- Cohort 2 (Experimental): HER2(+)&CLDN18.2(+)&PD-L1(-)
  Interventions: Drug: Trastuzumab; Drug: S-1; Drug: SHR-A1904
- Cohort 3 (Experimental): HER2(2+ or 3+)&CLDN18.2(-)&PD-L1(-)
  Interventions: Drug: S-1; Drug: SHR-A1811
- Cohort 4 (Experimental): HER2(-)&CLDN18.2(+)&PD-L1(+)
  Interventions: Drug: Adebrelimab; Drug: S-1; Drug: SHR-A1904
- Cohort 5 (Experimental): HER2(-)&CLDN18.2(-)&PD-L1(+)
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Drug: SHR-1701
- Cohort 6 (Experimental): HER2(-)&CLDN18.2(+)&PD-L1(-)
  Interventions: Drug: S-1; Drug: SHR-A1904
- Cohort 7 (Experimental): HER2(-)&CLDN18.2(-)&PD-L1(-)
  Interventions: Drug: Apatinib; Drug: S-1; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Trastuzumab — iv，d1
  Arms: Cohort 1; Cohort 2
Drug: Adebrelimab — iv，d1，q3w
  Arms: Cohort 1; Cohort 4
Drug: Apatinib — po，qd，d1-21，q3w
  Arms: Cohort 7
Drug: S-1 — po，bid，d1-14，q3w
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 6; Cohort 7
Drug: Capecitabine — po，bid，d1-14
  Arms: Cohort 5
Drug: Oxaliplatin — iv，d1，q3w
  Arms: Cohort 5; Cohort 7
Drug: zolbetuximab — iv，d1
  Arms: Cohort 1
Drug: SHR-A1811 — iv，d1 ，q3w
  Arms: Cohort 3
Drug: SHR-A1904 — iv，d1 ，q3w
  Arms: Cohort 1; Cohort 2; Cohort 4; Cohort 6
Drug: SHR-1701 — iv，d1 ，q3w
  Arms: Cohort 5

SUMMARY:
This study is a prospective, umbrella-design, Phase II clinical trial. Eligible participants with advanced or metastatic gastric cancer who are treatment-naïve for advanced-stage systemic therapy will undergo biomarker profiling (HER2, CLDN18.2, and PD-L1) via next-generation sequencing (NGS) or immunohistochemistry (IHC). Participants will be stratified into distinct molecular subtypes and assigned subtype-specific therapeutic regimens. The primary objectives are to assess treatment efficacy (e.g., objective response rate) and safety profiles across molecularly defined cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, regardless of gender;
2. Histologically or pathologically confirmed gastric adenocarcinoma or adenocarcinoma of the gastroesophageal junction;
3. Advanced or metastatic disease with no prior systemic therapy for advanced-stage disease (Patients who relapsed >6 months after completing neoadjuvant/adjuvant therapy are eligible, with prior neoadjuvant/adjuvant regimens not counted as prior lines of therapy);
4. At least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST v1.1);
5. Archival or fresh tumor tissue sample available for biomarker testing (HER2, CLDN18.2, and PD-L1 expression);
6. ECOG performance status: 0-1;
7. Life expectancy ≥12 weeks;
8. Adequate organ and bone marrow function meeting the following criteria:

   1. Hemoglobin ≥90 g/L (no blood transfusion within 14 days);
   2. Absolute neutrophil count (ANC) ≥1.5×10⁹/L;
   3. Platelet count ≥90×10⁹/L;
   4. Total bilirubin ≤1.5×upper limit of normal (ULN);
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN (≤5×ULN if liver metastases are present);
   6. Serum creatinine ≤1.5×ULN;
   7. Left ventricular ejection fraction (LVEF) ≥50% by echocardiography; QTc interval <450 ms for males and <470 ms for females;
9. Coagulation parameters:
10. For patients not on anticoagulation therapy: INR ≤1.5 and activated partial thromboplastin time (APTT) ≤1.5×ULN;
11. For patients receiving full-dose or parenteral anticoagulation: Stable anticoagulant dose for ≥2 weeks prior to enrollment, with coagulation tests within the therapeutic range;
12. Contraception requirements:
13. Women of childbearing potential must have a negative pregnancy test (serum or urine) within 14 days prior to enrollment and agree to use effective contraception during the study and for 3 months after the last dose;
14. Men must be surgically sterile or agree to use effective contraception during the study and for 3 months after the last dose;
15. Recovery from prior therapy-related toxicities to ≤Grade 1 (surgical wounds must be fully healed if applicable);
16. Voluntary participation with signed informed consent form and anticipated adherence to protocol requirements.

Exclusion Criteria:

1. History of gastrointestinal perforation and/or fistula within 6 months prior to treatment, or active gastrointestinal bleeding within 3 months;
2. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage;
3. Known history of hypersensitivity to any component of the investigational drug(s) or excipients;
4. Prior treatments meeting any of the following:

   1. Received any investigational drug within 4 weeks prior to the first dose of the study drug or within 5 half-lives of the last investigational agent (whichever is shorter);
   2. Concurrent enrollment in another interventional clinical study (observational or follow-up studies are permitted);
   3. Received antitumor therapy (including radiotherapy, chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologics, or tumor embolization) within 2 weeks prior to the first dose of the study drug;
5. History of leptomeningeal metastasis or current active brain metastases;
6. Severe infection (CTCAE v5.0 Grade >2) within 4 weeks prior to the first dose of the study drug (e.g., pneumonia requiring hospitalization, bacteremia, or septic complications); active pulmonary inflammation on baseline chest imaging, or signs/symptoms of infection requiring oral/IV antibiotics within 2 weeks prior to the first dose (prophylactic antibiotics excluded);
7. History of interstitial lung disease (except radiation pneumonitis without steroid treatment or non-infectious pneumonitis);
8. Active tuberculosis (TB) infection confirmed by medical history or CT scan, history of active TB within 1 year prior to enrollment, or untreated active TB diagnosed >1 year prior to enrollment;
9. Diagnosis of another malignancy within 5 years prior to the first dose of the study drug, except malignancies with low metastatic/lethal risk (5-year survival rate >90%), such as adequately treated basal cell carcinoma, squamous cell skin cancer, or carcinoma in situ of the cervix;
10. Pregnant or lactating women;
11. Other conditions deemed by the investigator to jeopardize subject safety or trial integrity, including severe comorbidities (e.g., psychiatric disorders), clinically significant laboratory abnormalities, or social/family factors that may compromise protocol adherence or data collection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2029-08-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 2year
  Objective Response Rate (ORR) is defined as the proportion of patients who achieve a complete response (CR) or partial response (PR) to a therapeutic intervention, as assessed by standardized criteria (e.g., RECIST 1.1 for solid tumors). It serves as a key efficacy endpoint in early-phase clinical trials to evaluate the preliminary antitumor activity of investigational therapies.

SECONDARY OUTCOMES:
OS | 2year
  Overall Survival (OS) is defined as the time from randomization (or initiation of treatment) until death from any cause. It is considered the gold standard endpoint in oncology clinical trials due to its objectivity and direct relevance to patient benefit.